CLINICAL TRIAL: NCT04009070
Title: Effect of Acupuncture on Nausea, Vomiting, Pain, PGE2 and IL 6 in Septorhinoplasty Operations; Prospective, Randomized, Controlled Study
Brief Title: Effect of Acupuncture on Nausea, Vomiting, Pain, PGE2 and IL 6 in Septorhinoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yavuz Orak, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2018/12-17
Record Dates: First submitted 2019-03-08; First posted 2019-07-05 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Pain; Acupuncture
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Group A: Acupuncture Group Group C: Control Group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Active Comparator): Group A: Acupuncture group:Group A: Acupunctur will be applied to the Acupunctur group 24 hours prior to bilateral PC6 (approximately two cm above the midline of the wrist line) and ST 36 (approximately 1-2 cm laterally on the tibia) . The tape (Needle Press) will stay for 24 hours.
  Needle Press: Pres Needle: 0.22x1.5 mm needle
  Interventions: Device: Acupuncture Pres Needle: 0.22x1.5 mm needle
- Control Group (No Intervention): Group C: Control group

INTERVENTIONS:
Device: Acupuncture Pres Needle: 0.22x1.5 mm needle — Acupunctur group; Acupunctur preoperatively 24 hours before bilateral PC6 (approximately two cm above the midline of the wrist line) and ST 36 (approximately 1-2 cm laterally from the tuberocyte tibia). The tape (Needle Press) will remain for 24 hours after surgery.
  Arms: Acupuncture

SUMMARY:
Acupuncture has emerged in China about 2,000 years ago and is one of the oldest medical procedures in the world.Later acupuncture was introduced to other regions such as Asia, Europe and the United States.The most extensive use of acupuncture is for pain relief.Especially, postoperative nausea and vomiting have been studied.In one study, PC6 (approximately two cm above the midline of the wrist line) showed antiemetic effect, with the addition of other acupuncture points, it proved to have a protective effect in the treatment of postoperative nausea and vomiting.ST36 (Approximately 1-2 cm laterally from the tuberocyte tibia) is an acupuncture point used in the treatment of diseases such as inflammation, acute pain, hypertension and gastrointestinal disorders.

DETAILED DESCRIPTION:
Patients will be determined as Group A: Acukupuncture group and Group C as Control group and 35 patients will be included in the study. Both groups will be given an intravenous (i.v) route in the preoperative patient room, PGE2, IL 6 will be taken for blood and 0.09% NaCl will be started. Group A preoperatively, 24 hours prior to bilateral PC6 (approximately two cm above the midline of the wrist line) and ST 36 (approximately 1-2 cm laterally from the Tibia) to be applied to the press needle (0.22x1.3 mm) and the tape (Needle Press will remain for 24 hours after surgery. Electrocardiography (ECG), noninvasive blood pressure (SBP-DBP), and peripheral arterial oxygen saturation (SpO2) monitoring will be applied to the patients. In the induction of anesthesia, Pentotal 5 mg / kg, Fentanyl 0.5 mcg / kg, and rocuronium 0.6 mg / kg will be used. Anesthesia maintenance will be provided with a 2% concentration of sevoflurane, 50% nitrous oxide (N2O) and 50% oxygen (O2) mixture and appropriately intubated. Patients will be recorded with systolic blood pressure (SBP), diastolic blood pressure (heart failure), heart rate (HR), mean arterial pressure (MAP) and SpO2, 5, 15, 30, 60, 120 minutes (min) after induction.

Patients in Group A and Group C had a saturation value of 97% or more, and exhaled if breathing effort was sufficient. Atropine and neostigmine will be used to neutralize muscle relaxants. Contramal 1mg / kg will be applied to the patients as standard by 20 minutes before the end of surgery. Following the termination of the surgical intervention, the anesthesia gases will be cut and 100% O2 will be inhaled with the mask until all the cases are compiled. 5.dk follow-up and extubation period of the patients will be taken to the postoperative rest room after being followed up on the operating table. 30. Min follow-up will be sent to their services after being done here. Postoperative 60 min, 3 h, 6 h, 12 h, 24 h, sore throat, nausea, vomiting, cough, itching, dysphagia, sore throat and analgesic needs, whether pain, assessment will be made. VAS score will be used to evaluate pain. Paracetamol will be applied to all patients when analgesia needs. At 24 hours postoperatively, blood will be taken to look for PGE2 and IL6 values.Preoperative and postoperative PGE2 and IL 6 values will be compared between the groups of the acupuncture group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II group
* Aged 18-75
* Volunteer to participate in the study
* Conscious patients.

Exclusion Criteria:

* Not wanting to participate
* Unconscious
* Having a hearing and speech problem
* Allergic disease and bleeding disorder
* Respiratory problems

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change Pain Scores | 5 minute,30 minute, 60 minute, 3 hours, 6 hours, 12 hours, 24 hours after the operation
  VAS (Visual analog scale) Score. from 1 to 10 , 0: No pain, 10: 10 pain that can not be tolerated
PG E2 | Change from baseline and concentration of preoperativ and postoperative values at 24.hours
  To evaluate the impact on the circulating levels of PG E2 ng/ml
IL 6 | Change from baseline and concentration of preoperativ and postoperative values at 24.hours
  To evaluate the impact on the circulating levels of IL 6 ng/ml
Nause and Vomiting | After operation at 5 minutes, 30 minutes, 60 minutes,3 hours, 6 hours, 12 hours, 24 hours
  Yes or No Nause and vomiting

SECONDARY OUTCOMES:
Blood Pressure | During operation at 5 minute, 15 minutes, 30 minutes, 60 minutes, 120 minutes and After operation at 5 minutes, 30 minutes, 60 minutes,3 hours, 6 hours, 12 hours, 24 hours after operation
  Systolic blood pressue mmHg , diastolic blood pressure mmHg, mean arterial pressure mmHg,
Heart rate | During operation at 5 minute, 15 minutes, 30 minutes, 60 minutes, 120 minutes and After operation at 5 minutes, 30 minutes, 60 minutes,3 hours, 6 hours, 12 hours, 24 hours
  heart rate ,
Change of Itching, cough, sore throat, difficulty in swallowing | Do Patients have any Itching, cough, sore throat, difficulty in swallowing in 5 minute,30 minute, 60 minute, 3 hours, 6 hours, 12 hours, 24 hours after operation
  it will be asked if there are Itching, cough, sore throat, difficulty in swallowing.more in which group.
oxygen follow-up | at 5 minute, 15 minutes, 30 minutes, 60 minutes, 120 minutes during
  oxygen saturation
oxygen follow-up | 30 minutes, 60 minutes,3 hours, 6 hours, 12 hours, 24 hours after the operation,
  oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: yavuz orak, md, Principal Investigator — Kahramanmaraş Sutcu Imam University Faculty of Medicine
Locations (1):
- Kahramanmaras Sutcu Imam University Faculty of Medicine, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orak Y, Baylan FA, Bilgen F, Orak F, Ural A, Yildiz S, Sagiroglu S, Karaduman H, Doganer A. The Effect of Acupuncture on Pain, Prostaglandin E2, and Interleukin-6 in Septorhinoplasty Operations: A Randomized Clinical Trial. Anesthesiol Res Pract. 2025 Dec 7;2025:7816719. doi: 10.1155/anrp/7816719. eCollection 2025. PMID 41362812